CLINICAL TRIAL: NCT01170689
Title: The Prevalence of Obesity For Schizophrenia Inpatients in Taiwan
Status: Completed | Type: Observational
Sponsor: TsaoTun Psychiatric Center, Department of Health, Taiwan (Other)
Responsible Party: Han-Yi Ching, Psaotun psychiatric center,department of health
Other Study IDs: Tsao-Tun Psychiatric Center
Record Dates: First submitted 2010-07-26; First posted 2010-07-27 (Estimated); Last update posted 2010-07-28 (Estimated); Status verified 2010-07

CONDITIONS: Schizophrenia; Obesity
Keywords: Schizophrenia; inpatient; obesity; prevalence
MeSH Terms: conditions — Schizophrenia; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Inpatient schizophrenia or schizoaffective disorder

SUMMARY:
This study is the first hospital-based, cross-sectional study to discuss the prevalence of obesity among 710 inpatients with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis as ICD 295
2. Living in rehabilitation ward during 2010/03/22~2010/04/02

Exclusion Criteria:

none

Ages: 20 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 710 adult schizophrenia patients living in the chronic ward in Tsau-Tun psychiatric center during the first week in March 2010
Sampling Method: Probability Sample
Enrollment: 710 (Actual)
Dates: Start 2010-03; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Body mass index (BMI) | cross-sectional study, check one time

SECONDARY OUTCOMES:
waist circumference | cross-sectional study, check for one time

CONTACTS AND LOCATIONS:
Overall Officials: Ching Han-Yi, MD, Principal Investigator — Tsaotun Psychiatric Center
Locations (1):
- Tsao-Tun Psychiatric Center, Nantou City, Taiwan